CLINICAL TRIAL: NCT07169175
Title: A Multicenter, Open-label, Single-arm, Dose Escalation and Expansion, Phase I/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SNUG01 in Adult Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Phase Ⅰ/Ⅱa Study of SNUG01 in Adult Subjects With ALS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SineuGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNUG01-101
Record Dates: First submitted 2025-08-08; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3 Ascending Dose Levels, Single Injection by Intrathecal(IT) (Experimental)
  Interventions: Drug: SNUG01

INTERVENTIONS:
Drug: SNUG01 — AAV (adeno-associated virus) Gene therapy

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and preliminary efficacy of SNUG01 in in adult subjects with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
This is a 52-week, multicenter, open-label, single-arm, dose escalation and expansion Phase Ⅰ/Ⅱa study of SNUG01 in adults with ALS. Safety will be the primary focus, with secondary emphasis on immunogenicity, PK and preliminary clinical efficacy of SNUG01.

ELIGIBILITY:
* Key Inclusion Criteria**:

  * Subjects who are able to provide written informed consent form (ICF).
  * Subjects who are males or females must be ≥ 18 years and ≤ 80 years of age at the screening visit.
  * Subjects who have clinically definite ALS, clinically probable ALS, or clinically probable-laboratory supported ALS as specified in the revised version of the El Escorial World Federation of Neurology criteria.
  * Subjects must have an ALS disease duration (from first symptom onset to the screening visit) ≤ 2 years.
  * Subjects with a body mass index (BMI) ≥ 19 kg/m2 at the screening visit.
  * Subjects whose percent-predicted Forced Vital Capacity (%FVC) is ≥ 70% or percent-predicted Slow Vital Capacity (%SVC) is ≥ 60%, adjusted for sex, age, and height at the screening visit.
  * The ALSFRS-R score ≥ 30 during the screening period, and the three respiratory scores (dyspnea, upright respiration, and respiratory insufficiency) must be full marks.
* Key Exclusion Criteria**:

  * Serum Anti-AAV9 neutralizing antibody titer ≥ 1:100.
  * Current or previous exposure to gene therapy, stem cell products, and solid organ transplantation.
  * Subjects who have implanted or are estimated to require a diaphragmatic pacing system during the study period.
  * Any thromboembolic event, such as deep vein thrombosis, pulmonary arteriovenous embolism, and jugular vein embolism, has occurred within 6 months before the administration.
  * Suffering from autoimmune diseases or ongoing immune-related therapy, except intranasal, inhalation, ocular, topical, intra-articular corticosteroid therapy or corticosteroid physiological replacement therapy.
  * Active or chronic uncontrolled infection within 4 weeks before the administration, deemed unacceptable in the discretion of the investigator.
  * Evidence of human immunodeficiency virus (HIV) and treponema pallidum (TP) infection, as documented by the treatment for HIV or TP, or by HIV or TP antibodies positivity at the screening visit.
  * Has a positive serum pregnancy test at screening (females of childbearing potential only), a positive urine or serum pregnancy test at baseline (Day -1. females of childbearing potential only), or is nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of SNUG01 administered by intrathecal. | up to 1 year after administration
  Dose-limiting toxicity (DLT), adverse events (AEs), clinically significant changes in vital signs, physical examination, clinical laboratory tests (hematology, biochemistry, urinalysis, coagulation, cardiac enzymes, etc.) and 12-lead ECG, etc.
To recommend the optimal expansion dose of SNUG01 that demonstrates acceptable safety with maximum preliminary efficacy administered by IT. | up to 1 years

SECONDARY OUTCOMES:
Immunogenicity of SNUG01 | up to 1 years
  Change of anti-SG001 antibody and anti-AAV9 neutralizing antibody in serum, change of anti-AAV9 neutralizing antibody in CSF.
PK of SNUG01 (Biodistribution and Viral Shedding) | up to 1 years
  SG001 protein level in CSF, viral vector DNA in serum, viral shedding in saliva, urine, and feces.
Preliminary Clinical Efficacy of SNUG01 | up to 1 years
  Change in the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) , the Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) , the percent-predicted Forced Vital Capacity (%FVC) / percent-predicted Slow Vital Capacity (%SVC) and muscle strength, the Patient Health Questionnaire (PHQ-9) and NfL level in CSF and serum from baseline to Week 48 after administration.

CONTACTS AND LOCATIONS:
Locations (4):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- China (3):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang